CLINICAL TRIAL: NCT03796767
Title: Salvage Oligometastasectomy and Radiation Therapy in Recurrent Prostate Cancer (SOAR)
Brief Title: Salvage Oligometastasectomy and Radiation Therapy in Recurrent Prostate Cancer
Acronym: SOAR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI115811; NCI-2018-03418 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Prostate Carcinoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Malignant Neoplasm in the Lymph Nodes; Oligometastasis; Prostate Adenocarcinoma; PSA Failure
MeSH Terms: conditions — Prostatic Neoplasms; Lymphatic Metastasis | interventions — Radiation Dose Hypofractionation; Radiotherapy, Intensity-Modulated; Metastasectomy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (radiation therapy) (Experimental): Patients with bone metastases undergo SBR) or hypofractionated radiation per institutional standard of care guidelines at investigator's discretion.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy
- Arm B (salvage oligometastasectomy) (Experimental): Patients with nodal metastases undergo salvage oligometastasectomy.
  Interventions: Procedure: Metastasectomy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm C (salvage oligometastasectomy, radiation therapy) (Experimental): Patients with nodal metastases undergo salvage oligometastasectomy. Following recovery, patients undergo SBRT or hypofractionated radiation per institutional standard of care guidelines at investigator's discretion. Within 4 months following completion of salvage therapy (defined as the combination of oligometastasectomy and/or bone radiation) and depending on PSA response as well as previous treatment, patients may receive adjuvant nodal IMRT.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Metastasectomy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation
  Arms: Arm A (radiation therapy); Arm C (salvage oligometastasectomy, radiation therapy)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
  Arms: Arm C (salvage oligometastasectomy, radiation therapy)
Procedure: Metastasectomy — Undergo salvage oligometastasectomy
  Arms: Arm B (salvage oligometastasectomy); Arm C (salvage oligometastasectomy, radiation therapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Arm A (radiation therapy); Arm C (salvage oligometastasectomy, radiation therapy)

SUMMARY:
This phase II trial studies how well surgery and radiation therapy work in treating patients with prostate cancer that has come back or spread to other parts of the body. Radiation therapy uses high energy beams to kill tumor cells and shrink tumors. Surgical procedures, such as oligometastasectomy, may remove tumor cells that have spread to other parts of the body. Surgery and radiation therapy may work better in treating patients with prostate cancer that has come back or spread to other parts of the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess response to treatment of oligometastatic disease.

SECONDARY OBJECTIVES:

I. To assess additional measurements of response to treatment of oligometastatic disease.

II. To assess prostate-specific antigen (PSA) progression free-survival following treatment of oligometastatic disease.

III. To assess time to disease recurrence following treatment of oligometastatic disease.

IV. To assess time to initiation of antiandrogen therapy (ADT) for metastatic prostate cancer following treatment of oligometastatic disease.

V. To assess the rate of undetectable PSA following treatment of oligometastatic disease in subjects who have previously undergone prostatectomy.

VI. To assess safety. VII. To assess the impact of study treatment on change in quality of life over three years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate.
* Recurrent prostate carcinoma after definitive therapy for primary disease defined as:

  * Post-prostatectomy (with/without adjuvant radiotherapy): Patients must have a detectable or rising PSA level that is > 0.05 ng/mL, with a second confirmatory level of > 0.05 ng/mL after a minimum of 1 week.
  * Post radiotherapy/ablation (without radical prostatectomy): PSA rise >= 2ng/mL over nadir.
* Subjects treated with prior definitive radiotherapy for prostate cancer who have positive molecular imaging (e.g., fluciclovine PET/CT scan or other per PI discretion) suggesting recurrent intraprostatic disease must undergo transrectal ultrasound (TRUS) biopsy less than or equal to one year before study enrollment:

  * If the TRUS biopsy is negative, no additional treatment is required to the prostate in addition to that of scan positive sites.
  * If the TRUS biopsy is positive, subject must undergo salvage prostatectomy or salvage radiotherapy to the primary site concurrently with the study treatment per the treatment protocol algorithm.
  * NOTE: Biopsy is not required for prostate fossa recurrences after radical prostatectomy.
* Oligometastatic disease defined as 10 or fewer metastatic lesions to lymph nodes and/or bones only.
* For patients with oligometastatic disease involving lymph nodes, metastasis is confined to the pelvic or para-aortic (below IMA) regions on molecular imaging (e.g., fluciclovine PET/CT or PSMA PET/CT scan or other per PI discretion).
* All subjects must be surgical candidates if surgery is indicated per the treatment algorithm.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
* Use of condoms for male subjects who have not had surgical removal of their prostate and have a partner of child bearing potential beginning at the time of informed consent form (ICF) signature and lasting until at least 6 months after the last radiation treatment. Because of the potential side effect on spermatogenesis associated with radiation, female partners of childbearing potential must agree to use a highly effective contraceptive method during and for 6 months after completing treatment.
* Recovery to baseline or =< grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v)5 from toxicities related to any prior treatments, unless adverse event (AE)(s) are clinically non-significant and/or stable on supportive therapy as determined by the treating physician.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Known brain or visceral metastases other than lymph nodes as defined by CT, MRI, or othermolecular imaging (e.g., fluciclovine PET/CT or PSMA PET/CT scan or other per PI discretion).
* Patients actively receiving hormone therapy for prostate cancer. Patients may have received hormone therapy perviously but must have documented non-castrate levels of testosterone (>50 ng/dL)
* Prior or concurrent malignancy whose natural history or treatment, in the opinion of the enrolling investigator, may have the potential to interfere wih the safety or efficay assessment of the investigational treatment protocol of the study.
* Use of finasteride within 30 days prior to initiation of therapy. Baseline PSA should not be obtained prior to 30 days after stopping finasteride.
* Use of dutasteride within 90 days prior to initiation of therapy. Baseline PSA should not be obtained prior to 90 days after stopping dutasteride.
* Use of any prohibited therapy.
* Active, uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mmHg systolic or > 100 mmHg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis, pulmonary embolism) within 6 months before first dose.
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration or within 30 days of registration.
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Sanchez, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Radiation Therapy) | Arm B (Salvage Oligometastasectomy) | Arm C (Salvage Oligometastasectomy, Radiation Therapy)
Started | 2 | 18 | 0
Completed | 2 | 18 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Arm C.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Radiation Therapy) | Arm B (Salvage Oligometastasectomy) | Arm C (Salvage Oligometastasectomy, Radiation Therapy) | Total
Number analyzed (Participants) | 2 | 18 | 0 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 8 | 0 | 10
  >=65 years | 0 | 10 | 0 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.50 (0.71) | 66.50 (6.84) |  | 66.00 (6.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 2 | 18 | 0 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 1 | 17 | 0 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 17 | 0 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 18 |  | 20
Height [Mean (Standard Deviation); unit: cm] | 173.9 (5.39) | 177.78 (7.32) |  | 177.40 (7.13)
Weight [Mean (Standard Deviation); unit: kg] | 180.00 (11.31) | 93.02 (11.94) |  | 91.72 (12.26)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.35 (2.11) | 29.43 (3.27) |  | 29.12 (3.27)
PSA at Time of Initial Definitive Treatment [Mean (Standard Deviation); unit: ng/mL] — Prostate-Specific Antigen (PSA) is a protein produced by tissue in the prostate. An elevated PSA value can be a sign of prostate cancer.
  ng/mL | 9.80 (7.78) | 9.18 (14.01) |  | 9.24 (13.37)
Number of Nodal Lesions Present [Mean (Full Range); unit: Lesions] — Nodal lesions in prostate cancer are lymph nodes near the prostate that contain cancer cells.
  Lesions | 0 [0 to 0] | 2.06 [1 to 6] |  | 1.85 [0 to 6]
ECOG [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) is a common oncology metric used to describe a patient's level of functioning.
  Participants
    0 Fully active | 1 | 18 | 0 | 19
    1 Restricted | 1 | 0 | 0 | 1
    2 Ambulatory | 0 | 0 | 0 | 0
    3 Limited selfcare | 0 | 0 | 0 | 0
    4 Completely disabled | 0 | 0 | 0 | 0
    5 Dead | 0 | 0 | 0 | 0
Histology [Count of Participants; unit: Participants] — Adenocarcinoma of the prostate is a malignant tumor from the glands in the prostate.
  This will report patients who had histologically proven adenocarcinoma of the prostate only or of the prostate and secondary histology
  Participants
    Adenocarcinoma of the prostate | 2 | 18 | 0 | 20
    Adenocarcinoma of the prostate + secondary histology | 0 | 0 | 0 | 0
Total Gleason at Definitive Treatment [Count of Participants; unit: Participants] — Total Gleason scores are prostate cancer grading systems based on microscopy of tissue samples. Scores range from 6 to 10, with lower scores indicating lower grade cancer and higher scores indicating higher grade cancer.
  Participants
    6 | 0 | 1 | 0 | 1
    7 | 1 | 13 | 0 | 14
    8 | 1 | 1 | 0 | 2
    9 | 0 | 3 | 0 | 3
T Stage [Count of Participants; unit: Participants] — Measure Description: With the Tumor Node Metastasize (TNM) system, the T Stage describes the extent of the main tumor.
  T2: Organ confined T2a: Tumor spread to ≤ half of one side of the prostate T2b: Tumor spread to > half of one side of the prostate T2c: Tumor spread to both sides of the prostate T3: Extraprostatic extension T3a: Extraprostatic extension (unilateral or bilateral) or microscopic invasion of bladder neck T3b: Tumor invades seminal vesicle(s) T4: Tumor is fixed or invades adjacent structures other than seminal vesicles
  Participants
    T2 | 0 | 2 | 0 | 2
    T2a | 0 | 0 | 0 | 0
    T2b | 0 | 0 | 0 | 0
    T2c | 0 | 5 | 0 | 5
    T3 | 0 | 0 | 0 | 0
    T3a | 2 | 6 | 0 | 8
    T3b | 0 | 5 | 0 | 5
N Stage [Count of Participants; unit: Participants] — With the Tumor Node Metastasize (TNM) system, the N Stage describes if cancer spread to nearby lymph nodes.
  NX: Regional lymph nodes cannot be assessed N0: No positive regional nodes N1: Metastases in regional node(s)
  Participants
    NX (regional lymph nodes cannot be assessed) | 0 | 1 | 0 | 1
    N0 | 2 | 11 | 0 | 13
    N1 | 0 | 5 | 0 | 5
    Unknown / Not assessed | 0 | 1 | 0 | 1
M Stage [Count of Participants; unit: Participants] — With the Tumor Node Metastasize (TNM) system, the M Stage describes if cancer spread (metastasized) to other parts of the body.
  M0: No distant metastasis M1: Distant metastasis M1a: Nonregional lymph node(s) M1b: Bone(s) M1c: Other site(s) with or without bone disease
  Participants
    M0 | 2 | 6 | 0 | 8
    M1 | 0 | 0 | 0 | 0
    Unknown / Not assessed | 0 | 12 | 0 | 12
Overall Stage [Count of Participants; unit: Participants] — In the Tumor Node Metastasize (TNM) system, overall stage is the extent of cancer based on 5 items:
  1. Extent of the main tumor (T)
  2. If cancer spread to nearby lymph nodes (N)
  3. If cancer spread (metastasized) to other parts of the body (M)
  4. PSA level at diagnosis
  5. Grade Group (from Gleason score)
  Stage IIB (T1-2, N0, M0, PSA <20, Grade 2) Stage IIIA (T1-2, N0, M0, PSA >=20, Grade 1-4) Stage IIIB (T3-4, N0, M0, Any PSA, Grade 1-4) Stage IIIC (Any T, N0, M0, Any PSA, Grade 5) Stage IVA (Any T, N1, M0, Any PSA, Any Grade) Stage IVB (Any T, Any N, M1, Any PSA, Any Grade)
  Participants
    Stage IIB | 0 | 3 | 0 | 3
    Stage IIIA | 0 | 2 | 0 | 2
    Stage IIIB | 2 | 1 | 0 | 3
    Stage IIIC | 0 | 2 | 0 | 2
    Stage IVA | 0 | 2 | 0 | 2
    Stage IVB | 0 | 1 | 0 | 1
    Unknown / Not assessed | 0 | 7 | 0 | 7
Prior radiotherapy [Count of Participants; unit: Participants] — Radiotherapy (or Radiation therapy) is used to kill cancer cells and shrink tumors with high doses of radiation.
  Participants
    None | 0 | 11 | 0 | 11
    Definitive Radiotherapy - Prostate (should be salvage radiation - prostate) | 0 | 2 | 0 | 2
    Adjuvant/Salvage Radiotherapy - Prostate | 0 | 4 | 0 | 4
    Adjuvant/Salvage Radiotherapy - Pelvis + Prostate | 2 | 1 | 0 | 3
Prior exposer to Androgen deprivation therapy (ADT) [Count of Participants; unit: Participants] — ADT is a medication that reduces the amount of androgens in the body. This is used as a treatment for prostate cancer as androgens are important for prostate cancer cell growth. Hence, ADT can slow the cancer's progression.
  Participants
    Yes | 1 | 5 | 0 | 6
    No | 1 | 13 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Prostate-specific Antigen (PSA) ≥ 50% 6 Months After Completion of All Treatment
Description: The primary outcome measure will report the count of patients achieving a PSA decline >= 50% at 6 months after completion of treatment (salvage + - adjuvant).
  Prostate-Specific Antigen (PSA) is a protein produced by tissue in the prostate. An elevated PSA value can be a sign of prostate cancer.
Time Frame: 6 months after completion of 5-21 weeks of treatment
Population: No participants were enrolled in Arm C.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Radiation Therapy) | Arm B (Salvage Oligometastasectomy) | Arm C (Salvage Oligometastasectomy, Radiation Therapy)
Number analyzed (Participants) | 2 | 18 | 0
Participants
  Yes | 0 | 8 | 0
  No | 2 | 10 | 0

2. Secondary Outcome: Prostate-specific Antigen (PSA) ≥ 50% 12 Months After Completion of All Treatment
Description: Defined according to Prostate Cancer Working Group (PCWG3) criteria as the proportion of patients achieving a PSA decline >= 50% at 12 months after completion of treatment (salvage + - adjuvant).
  Prostate-Specific Antigen (PSA) is a protein produced by tissue in the prostate. An elevated PSA value can be a sign of prostate cancer.
Time Frame: 12 months after completion of 5-21 weeks of treatment
Population: No participant was enrolled on Arm C
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Radiation Therapy) | Arm B (Salvage Oligometastasectomy) | Arm C (Salvage Oligometastasectomy, Radiation Therapy)
Number analyzed (Participants) | 2 | 18 | 0
Participants
  Yes | 1 | 4 | 0
  No | 1 | 14 | 0

3. Secondary Outcome: Prostate-specific Antigen (PSA) ≥ 90%
Description: This outcome will report the count of patients achieving a PSA decline ≥ 90% 6 at 6 and12 months after completion of treatment (salvage + - adjuvant).
  Prostate-Specific Antigen (PSA) is a protein produced by tissue in the prostate. An elevated PSA value can be a sign of prostate cancer.
Time Frame: 6 and 12 months after completion of 5-21 weeks of treatment 6 Months After Completion of All Treatment6 Months After Completion of All Treatment
Population: No participants were enrolled in Arm C.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Radiation Therapy) | Arm B (Salvage Oligometastasectomy) | Arm C (Salvage Oligometastasectomy, Radiation Therapy)
Number analyzed (Participants) | 2 | 18 | 0
Participants
  PSA decline ≥ 90% at 6 Months: Yes | 0 | 5 | 0
  PSA decline ≥ 90% at 6 Months: No | 2 | 13 | 0
  PSA decline ≥ 90% at 12 Months: Yes | 0 | 4 | 0
  PSA decline ≥ 90% at 12 Months: No | 2 | 14 | 0

4. Secondary Outcome: PSA Progression Free-survival
Description: The proportion of subjects without PSA progression (defined using Prostate Cancer Working Group 3 Criteria PCWG3), evaluated every 3 months for 3 years after completion of all treatment (salvage and adjuvant therapy).
Time Frame: Time elapsed between study enrollment and first occurrence of confirmed radiographic disease progression, assessed up to 3 years
Reporting Status: Not Posted, anticipated posting 2026-04

5. Secondary Outcome: To Assess Time to Disease Recurrence Following Treatment of Oligometastatic Disease.
Description: The time from study enrollment until the date of confirmed radiographic disease progression as defined by RECIST 1.1 and PCWG3.
Time Frame: Time elapsed between study enrollment and confirmed radiographic disease progression, up to 3 years
Reporting Status: Not Posted, anticipated posting 2026-04

6. Secondary Outcome: To Assess Time to Initiation of ADT for Metastatic Prostate Cancer Following Treatment of Oligometastatic Disease.
Description: The time from study enrollment to the initiation of ADT
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2026-04

7. Secondary Outcome: Undetectable PSA
Description: This outcome measure will report the count of participants with undetectable PSA after 6 and 12 months following completion of treatment (salvage ± adjuvant). Undetectable PSA is defined as the number of patients ever treated with prostatectomy whose PSA remains ≤ 0.2 ng/mL.
Time Frame: 6 and 12 months after completion of 5-21 weeks of treatment
Population: No participants were enrolled in Arm C
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Radiation Therapy) | Arm B (Salvage Oligometastasectomy) | Arm C (Salvage Oligometastasectomy, Radiation Therapy)
Number analyzed (Participants) | 2 | 18 | 0
Participants
  PSA ≤ 0.2 at 6 months: Yes | 0 | 7 | 0
  PSA ≤ 0.2 at 6 months: No | 2 | 11 | 0
  PSA ≤ 0.2 at 12 months: Yes | 1 | 4 | 0
  PSA ≤ 0.2 at 12 months: No | 1 | 14 | 0

8. Secondary Outcome: Number of Participants With Adverse Events (AE) by Grade
Description: This outcome measure will assess the safety and tolerability of the study treatment.
  The severity of AEs was assessed using CTCAE v5.0 criteria, a 1-5 scale with higher numbers indicating greater severity. Grade 1 indicates "mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated" and Grade 5 indicates "death related to AE".
  This outcome measure will report the count of participants who experienced each AE grade. Subjects were monitored for adverse events from the start of treatment until 28 days after the last dose of the study drug.
  Adverse events were collected every three months for one year after treatment discontinuation.
Time Frame: Up to 12 months after completion of 5-21 weeks of treatment
Population: No participants were enrolled in Arm C.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Radiation Therapy) | Arm B (Salvage Oligometastasectomy) | Arm C (Salvage Oligometastasectomy, Radiation Therapy)
Number analyzed (Participants) | 2 | 18 | 0
Participants
  CTCAE Grade: 1 | 1 | 11 |
  CTCAE Grade: 2 | 1 | 3 |
  CTCAE Grade: 3 | 0 | 0 |
  CTCAE Grade: 4 | 0 | 0 |
  CTCAE Grade: 5 | 0 | 0 |

9. Secondary Outcome: Quality of Life (QOL) - The Functional Assessment of Cancer Therapy - Prostate (FACT-P)
Description: FACT-P is a QOL questionnaires administered at the Response Assessment Visit. FACT-P is used to assess the health-related QOL in prostate cancer. Patients indicate which symptoms/problems they've experienced during the past week, from 1 Not at All to 4 Very Much.
  The assessment was scored according to the "FACT-P Scoring Guidelines (Version 4)". Individual items that were "reverse items" (high value indicates poor QOL) were subtracted from 4; reverse and normal items were added to calculate each subscale. The higher the subscale the better the QOL. The subscales and score ranges are: Physical Well-Being (0-28), Social/ Family Well Being (0-28), Emotional Well-Being (0-24), Functional Well Being (0-28), and Prostate Cancer Subscale (0-48)
  This outcome will report the mean score and 95% confidence interval of each subscale.
Time Frame: up to 45 days after the initiation of study therapy
Population: 1 participant did not complete this assessment in Arm A. 10 participants did not complete this assessment in Arm B. No participants were enrolled in Arm C.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm A (Radiation Therapy) | Arm B (Salvage Oligometastasectomy) | Arm C (Salvage Oligometastasectomy, Radiation Therapy)
Number analyzed (Participants) | 1 | 8 | 0
units on a scale
  Physical Well-Being | 26 | 25.75 [24.59 to 26.91] |
  Social/ Family Well Being | 16 | 24.13 [21.89 to 26.36] |
  Emotional Well-Being | 16 | 19.88 [16.97 to 22.78] |
  Functional Well Being | 14 | 24.50 [21.61 to 27.39] |
  Prostate Cancer Subscale | 41 | 36.50 [32.87 to 40.13] |

10. Secondary Outcome: Quality of Life (QOL): Expanded Prostate Cancer Index Composite (EPIC-26)
Description: EPIC-26 is a Health Related Quality of Life (HRQOL) questionnaires assessing the disease-specific aspects of prostate cancer and its therapies. This questionnaire asks patients to rank symptoms from 1 More than once a day to 5 Rarely or never.
  EPOC-26 reports 5 subscales: Urinary Incontinence Score, Urinary Obstructive/ Irritative Score, Bowel Score, Sexual Score, and Urinary Incontinence Score. Multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
Time Frame: up to 45 days after initiation of study therapy
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm A (Radiation Therapy) | Arm B (Salvage Oligometastasectomy) | Arm C (Salvage Oligometastasectomy, Radiation Therapy)
Number analyzed (Participants) | 1 | 8 | 0
units on a scale
  EPIC-26: Urinary Incontinence Score | 46 | 65.22 [51.21 to 79.23] |
  EPIC-26: Urinary Obstructive/ Irritative Score | 75 | 86.72 [76.51 to 96.93] |
  EPIC-26: Bowel Score | 100 | 94.27 [89.17 to 99.37] |
  EPIC-26: Sexual Score | 34.67 | 42.67 [16.06 to 69.27] |
  EPIC-26: Urinary Incontinence Score EPIC-26: Hormonal Score | 70 | 94.38 [88.69 to 100.06] |

ADVERSE EVENTS:
Time Frame: Collection of adverse events began with the first study salvage treatment (surgery OR radiotherapy for bone metastases) and ended 1 year after the last study treatment (including palliative radiotherapy if applicable) or until a new cancer treatment was initiated, up to 1 year.
Description: No participants were enrolled in Arm C.
Arm/Group | Arm A (Radiation Therapy) | Arm B (Salvage Oligometastasectomy) | Arm C (Salvage Oligometastasectomy, Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/18 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/18 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 12/18 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Radiation Therapy) (N=2) | Arm B (Salvage Oligometastasectomy) (N=18) | Arm C (Salvage Oligometastasectomy, Radiation Therapy) (N=0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT03796767/Prot_SAP_000.pdf